CLINICAL TRIAL: NCT00005484
Title: Predictors of Hospital-Based Care in Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5000; R29HL048237 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-03

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To identify clinical predictors of episodes of hospital-based care in people with asthma.

DETAILED DESCRIPTION:
BACKGROUND:

This study was of great practical importance because asthma is a common condition (3-5 percent of the population) which has had a recent, unexplained rise in morbidity and mortality. Many previous epidemiological studies focused on predictors of hospitalization for people with asthma seen in the emergency room. These studies were of limited value for the practicing physician who sees the vast majority of patients with asthma.

Results from this study should, for the first time, enable a profile to be constructed of the high risk patient with asthma which includes identification of modifiable risk factors. These results can be used for physician and patient education programs as well as to target medical intervention.

DESIGN NARRATIVE:

The study developed a key piece of information needed for outpatient care of patients with asthma; a profile of patients at risk for severe, potentially life-threatening exacerbations of asthma. The experimental design was a prospective study of 800 patients with asthma drawn from a large, pre-paid health care plan. The key advantage of this population was that all the care occurred within the health plan. Characteristics identified included demographic factors, socioeconomic status; patient characteristics such as tobacco use, atopy, pattern of medication use, self-reporting of compliance/adherence, attitudes about asthma; historical assessment of indoor air quality; characteristics of asthma such as duration of asthma, lung function, and variation in asthma symptoms; and speciality of physician. The outcome measures were obtained over a three year period and included all episodes of hospital-based care including hospitalizations, emergency room visits, and urgency care clinic visits. Based on these data, models were developed which assigned relative risk to each of the independent variables. These models were validated in a subset of the population.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-04; Study Completion 1997-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Osborne — Oregon Health and Science University

REFERENCES:
- [Background] Osborne ML, Vollmer WM, Linton KL, Buist AS. Characteristics of patients with asthma within a large HMO: a comparison by age and gender. Am J Respir Crit Care Med. 1998 Jan;157(1):123-8. doi: 10.1164/ajrccm.157.1.9612063. PMID 9445289
- [Background] Emery NL, Vollmer WM, Buist AS, Osborne ML. Self-reported food reactions and their associations with asthma. West J Nurs Res. 1996 Dec;18(6):643-54. doi: 10.1177/019394599601800603. PMID 9000872
- [Background] Sippel JM, Pedula KL, Vollmer WM, Buist AS, Osborne ML. Associations of smoking with hospital-based care and quality of life in patients with obstructive airway disease. Chest. 1999 Mar;115(3):691-6. doi: 10.1378/chest.115.3.691. PMID 10084477
- [Background] Osborne ML, Vollmer WM, Pedula KL, Wilkins J, Buist AS, O'Hollaren M. Lack of correlation of symptoms with specialist-assessed long-term asthma severity. Chest. 1999 Jan;115(1):85-91. doi: 10.1378/chest.115.1.85. PMID 9925066